CLINICAL TRIAL: NCT02076815
Title: A Phase III Randomized, Multicenter, Double-blind, Active Controlled Study to Compare the Efficacy and Safety of Two Different Anagrelide Formulations in Patients With Essential Thrombocythemia (TEAM-ET 2.0)
Brief Title: Anagrelide Retard in Essential Thrombocythemia
Acronym: TEAM-ET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AOP Orphan Pharmaceuticals AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AOP18007; 2013-003410-41 (EudraCT Number)
Record Dates: First submitted 2014-02-13; First posted 2014-03-04 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Essential Thrombocythemia
Keywords: myeloproliferative neoplasm; essential thrombocythemia; high risk patients; anagrelide
MeSH Terms: conditions — Thrombocythemia, Essential; Myeloproliferative Disorders | interventions — anagrelide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anagrelide retard (Experimental): Anagrelide Retard prolonged-release formulation
  Interventions: Drug: Anagrelide retard
- Thromboreductin (Active Comparator): Anagrelide immediate release formulation
  Interventions: Drug: Thromboreductin

INTERVENTIONS:
Drug: Anagrelide retard — Overencapsulated tablets or matched placebo, twice daily, 2-12 weeks titration to achieve stable platelet count, followed by 4 more weeks
  Other Names: Anagrelide retard 2 mg film coated tablet; ANAT2
  Arms: Anagrelide retard
Drug: Thromboreductin — Overencapsulated capsule, twice daily, 2-12 weeks titration to achieve the stable platelet count, followed by 4 more weeks
  Other Names: Anagrelide 0.5 mg capsule; ANAC05
  Arms: Thromboreductin

SUMMARY:
The purpose of this study is determine whether Anagrelide Retard is non-inferior to anagrelide immediate release form in treatment of essential thrombocythemia.

Essential thrombocythemia (ET) is a myeloproliferative neoplasm characterised by a sustained increase in platelet counts above the normal value (> 450 x 109/L) and increased megakaryopoiesis in the bone marrow, without secondary causes of thrombocytosis.

Anagrelide hydrochloride selectively reduces platelet numbers by inhibiting megakaryocyte development and maturation in humans, without affecting other cell lineages.

Anagrelide Retard is a new, prolonged release (PR) tablet formulation of anagrelide developed by AOP Orphan Pharmaceuticals AG. The rationale for developing this new formulation is based on the assumption of having a better tolerability while maintaining an efficacy comparable to that of the immediate release formulation.

The effects of Anagrelide Retard and Thromboreductin® will be compared in terms of mean platelet count measured by a central laboratory/centralized method at 3 time points during the maintenance phase.

DETAILED DESCRIPTION:
This is a randomised, multicentre, double-blind, active controlled study to compare the efficacy and safety of two different anagrelide formulations in patients with high-risk essential thrombocythemia (ET).

100 patients, either Anagrelide-treated or Anagrelide-naïve, with an indication to receive Thromboreductin® treatment, will be randomized into one of the two investigational medicinal product (IMP) groups (Anagrelide Retard or Thromboreductin®). Treatment allocation will be balanced within stratum (treated/naive) and age classes by central randomization. Naive patients will start with dose level 2 of the IMPs (i.e., 1 mg Thromboreductin® or 2 mg Anagrelide Retard). Anagrelide-treated patients will be switched to the dose level which is closest to the pre-study anagrelide dose at study start. Dose modifications in the titration phase will be done on a weekly basis (up to a maximum of 12 weeks) until "stable platelet counts" on two consecutive visits is achieved.

The periods of the study participation per patient are as follows:

* Screening (up to 7 days prior to randomization), ending with randomization/first IMP dose (Baseline Visit)
* Titration period (weekly visits for up to 12 weeks): to achieve "stable platelet counts" on two consecutive measurements (i.e. weekly visits)
* Maintenance period (weekly visits for 4 weeks): primary endpoint relevant period. The maintenance period for a patient starts at the visit with the second successive platelet count ≤400 G/L (or <600 G/L, if the dose cannot be increased any more due to intolerance or because the maximal dose allowed has already been reached) if the second platelet value measured lies in the range within ± 30% of the value measured at the previous visit.
* End of study (EoS) safety follow-up visit (28 days after the last maintenance visit/EoT for early termination).

ELIGIBILITY:
Inclusion Criteria:

* willing and able to give written informed consent prior to any study specific procedures and able to comply with the trial protocol
* confirmed diagnosis of ET according to 2008 WHO diagnostic criteria* (Swerdlow et al, 2008), defined as meeting all four criteria
* at high risk of experiencing ET-related events, indicated for Thromboreductin® treatment as defined by one or more of the following criteria: age ≥ 60 years, platelet counts ≥ 1000 G/L, increase of platelet count ≥ 300 G/L within 3 months, severe thrombohemorrhagic or ischemic symptoms in anamnesis
* either currently treated with anagrelide
* or ET treatment naive
* or anagrelide naive

Exclusion Criteria:

* Diagnosis of any myeloproliferative disorder other than ET
* Any known cause for a secondary thrombocytosis
* ET currently well controlled by another cytoreductive treatment than Anagrelide and the opportunity to continue to receive this treatment
* ET currently treated with combination of any two of the following agents: anagrelide, hydroxyurea, interferons, busulfan
* Hypersensitivity to either active or non-active ingredients of anagrelide or to any other excipients of the investigational products
* Known hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
* Cardiovascular disease grade 3 with a negative benefit/risk assessment or grade 4 (South West Oncology Group; Green and Weiss, 1992)
* Clinically significant abnormal laboratory values (excluding markers for ET) in investigator's opinion
* Severe renal insufficiency (creatinine clearance <30 ml/min)
* Moderate to severe hepatic insufficiency (ALT or AST > 5 times upper normal limit [UNL])
* White blood count (WBC) ≥ 15 G/L at screening
* Diagnosis of any malignancy, other than ET (except basal cell and squamous cell carcinomas of the skin and carcinoma in situ of the cervix that have been completely excised and are considered cured), within the last 3 years, or coexisting malignant, systemic disease
* Poorly controlled diabetes mellitus
* Known infection with hepatitis B, hepatitis C or HIV
* Pregnant or lactating women
* Women of childbearing potential or male patients, who have sexual intercourse with females of childbearing potential, not willing to use an effective method of contraception during the study.
* History of drug/alcohol abuse within the previous 2 years
* Participation in another investigational study within 4 weeks prior to informed consent signed or for a longer duration if specified in local regulations
* Any significant psychiatric disorder that, in the opinion of the investigator, might prohibit the understanding and giving of informed consent, or that might prevent the patient from completing the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Platelet count | weeks 13-17
  Mean value from three measurements

SECONDARY OUTCOMES:
platelet response | weeks 13-17
Time from randomization to entering maintenance period | up to 12 weeks
Study drug administration | weeks 1-17
Change in platelet counts in the titration period | baseline, week 12
Time from randomization until withdrawal | up to 17 weeks
Incidence, causality and intensity of adverse events | weeks 0-21
Incidence, intensity and outcomes of events leading to dose reduction or temporary or permanent treatment discontinuation | weeks 1-18
Need of medications to treat adverse events | weeks 0-21
ECG abnormalities | weeks 0-18
Ejection fraction | baseline, week 17, week 21
ECHO normal/abnormal | baseline, week 17, week 21

OTHER OUTCOMES:
Quality of Life | at week 1 and week 13
Plasma anagrelide concentration | At week 13, 15 and 17
Plasma anagrelide concentration | 1 min prior study treatment intake (morning dose), and 0.5, 1, 2, 3, 4, 6, 8, 10,12 (followed by evening dose), 13, 14, 15, 16, 18, 20, 24 hours after study treatment intake (morning dose)

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Gisslinger, Prof., MD, Principal Investigator — Vienna Medical University
Locations (19):
- Austria (3):
  - AOP Orphan Investigational Site Austria 2, Linz
  - AOP Orphan Investigational Site Austria 1, Vienna
  - AOP Orphan Investigational Site Austria 3, Wels
- Bulgaria (2):
  - AOP Orphan Investigational Site Bulgaria 1, Pleven
  - AOP Orphan Investigational Site Bulgaria 2, Sofia
- Lithuania (2):
  - AOP Orphan Investigational Site Lithuania 1, Kaunas
  - AOP Orphan Investigational Site Lithuania 2, Klaipėda
- Poland (6):
  - AOP Orphan Investigational Site Poland 5, Bialystok
  - AOP Orphan Insvestigational Site Poland 6, Gdansk
  - AOP Orphan Investigational Site Poland 4, Katowice
  - AOP Orphan Investigational Site Poland 3, Lublin
  - AOP Orphan Investigational Site Poland 2, Torun
  - AOP Orphan Investigational Site Poland 1, Warsaw
- Russia (6):
  - AOP Orphan Investigational Site Russia 1, Moscow
  - AOP Orphan Investigational Site Russia 2, Saint Petersburg
  - AOP Orphan Investigational Site Russia 5, Saint Petersburg
  - AOP Orphan Investigational Site Russia 4, Saint Petersburg
  - AOP Orphan Investigational Site Russia 6, Volgograd
  - AOP Orphan Investigational Site Russia 3, Yaroslavl